CLINICAL TRIAL: NCT03265340
Title: Clinical Effect of Deep Transcranial Magnetic Stimulation (dTMS) in Three Different Doses for the Treatment of Major Depressive Disorder
Brief Title: Clinical Effect of dTMS in Major Depressive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Section for Affective Disorders; Northern Stockholm Psychiatry (Other)
Responsible Party: Principal Investigator, Johan Lundberg, Section head, associate professor, MD PhD, Section for Affective Disorders; Northern Stockholm Psychiatry
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: dTMS dos-respons studie
Record Dates: First submitted 2016-10-28; First posted 2017-08-29 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: MAjor Depressive Disorder
Keywords: Transcranial Magnetic Stimulation
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Active Comparator): dTMS standard protocol 10 min session
  Interventions: Device: dTMS
- B (Active Comparator): dTMS standard protocol 20 min session
  Interventions: Device: dTMS
- C (Active Comparator): dTMS standard protocol 40 min session
  Interventions: Device: dTMS

INTERVENTIONS:
Device: dTMS

SUMMARY:
Aim: To test if there is a relation between deep Transcranial Magnetic Stimulation (dTMS) dose and clinical effect on Major Depressive Disorder (MDD) Method: 30 patients with moderate to severe MDD without concurrent medication will be randomised to three different treatment protocols of dTMS. Symptom severity of MDD will be quantified before, during and after dTMS.

DETAILED DESCRIPTION:
population: inclusion criteria:

1. Ongoing episode of MDD (ICD10 F32.x) according to MINI/SCID1.
2. Montgomery Asberg Depression Rating Scale (MADRS) score 20-60
3. TMS safe exclusion criteria:

1. Bipolar disorder 2. Substance abuse 3. fluoxetine treatment last three weeks 4. Other major Central Nervous System (CNS) disorder 5. Acute medical disorders 6. previous TMS or Electro Convulsive Treatment (ECT) <2 months before inclusion

ratings: MADRS at inclusion, baseline, weekly, at last visit Clinical Global Impression Severity (CGI-S) score at baseline, at last visit Global Self-Evaluation-Memory (GSE-My) at last visit Alcohol Use Disorder Identification Test (AUDIT-C) at inclusion EuroQual 5 Dimension (EQ5D) at baseline, at last visit Quick Inventory of Depressive Symptomatology Self Rating (QIDS-SR) baseline, weekly, last visit

condition: Each subject is randomised to condition A, B or C of dTMS (Brainsway): half the standard protocol (10 min; A), standard protocol (20 min; B) or double standard protocol (40 min, C). 20 treatment sessions/subject. 10 subjects in each group.

Primary endpoint: MADRS at baseline - MADRS at last visit (Intention TO Treat (ITT), Last Observation Carried Forward (LOCF))

ELIGIBILITY:
Inclusion Criteria:

* see above

Exclusion Criteria:

* see above

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Montgomery Asberg Depression Rating Scale (MADRS) score | baseline to last visit (treatment session 20, an average of four weeks)
  MADRS baseline - MADRS last visit (treatment session 20)

SECONDARY OUTCOMES:
Clinical Global Impression Severity (CGI-S) | baseline to last visit (treatment session 20, an average of four weeks)
  CGI-Sbaseline - CGI-S last visit (treatment session 20)
Montgomery Asberg Depression Rating Scale (MADRS) response | last visit (treatment session 20, an average of four weeks)
  fraction of subjects with >50% decrease in MADRS
Montgomery Asberg Depression Rating Scale (MADRS) remission | last visit (treatment session 20, an average of four weeks)
  fraction of subjects with MADRS <10 points
memory objective | baseline to last visit (treatment session 20, an average of four weeks)
  CPRS memory item at baseline - CPRS memory item at last visit
memory subjective | last visit (treatment session 20, an average of four weeks)
  GSE-my at last visit
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | baseline to last visit (treatment session 20, an average of four weeks)
  systematic safety evaluation and registration of side effects

CONTACTS AND LOCATIONS:
Overall Officials: johan lundberg, MD PhD, Principal Investigator — Norra Stockholms Psykiatri and Karolinska Institutet
Locations (1):
- Norra Stockholms Psykiatri, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No